CLINICAL TRIAL: NCT03961399
Title: Postmarketing, Prospective, Multicenter, Randomized and Blinded Study to Evaluate the Superior Efficacy of Cardiac Resynchronization Using the SyncAVTM Algorithm
Brief Title: Study to Evaluate the Superior Efficacy of Cardiac Resynchronization (SyncAVTM) Using the SyncAVTM Algorithm
Acronym: CRUSTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRUSTY
Record Dates: First submitted 2019-03-29; First posted 2019-05-23 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biventricular stimulation (BiV) group (Active Comparator): patients with Abbott Medical® CRT implanted with only biventricular stimulation (BiV).
  Interventions: Device: Abbott Medical® CRT device with biventricular stimulation (BiV)
- SyncAVTM stimulation group (Experimental): patients with Abbott Medical® CRT implanted and SyncAVTM stimulation activated
  Interventions: Device: Abbott Medical® CRT device with SyncAVTM stimulation function

INTERVENTIONS:
Device: Abbott Medical® CRT device with SyncAVTM stimulation function — patients with Abbott Medical® CRT device will be randomized and SyncAVTM stimulation will be activated.
  Arms: SyncAVTM stimulation group
Device: Abbott Medical® CRT device with biventricular stimulation (BiV) — patients with Abbott Medical® CRT device will be randomized and biventricular (BiV) stimulation will be activated.
  Arms: biventricular stimulation (BiV) group

SUMMARY:
Heart Failure (HF) is a cardiovascular disease secondary to a structural and / or functional alteration of the heart that prevents its correct function.

The Cardiac resynchronization therapy (CRT) aims to restore atrioventricular, inter and intraventricular synchrony in patients with systolic HF and wide depolarization of the ventricles (QRS). Although CRT has been shown to be effective, the rate of non-responders is high (30-50%).

One of the proposed reasons for the lack of response to the CRT is the lack of intrinsic conduction, since most of the time CRT is administered using biventricular stimulation (BiV). One of the limitations to achieve ventricular fusion are the dynamic physiological variations of the auriculo-ventricular (AV) interval.

The SyncAVTM algorithm is a new dynamic algorithm that manages to adjust the AV intervals outside the clinic.

The design of the present clinical study is post-marketing, prospective, multicenter, randomized and blind for the patient and the central echocardiography laboratory.

The objective of this study is to assess whether CRT with ventricular stimulation with fusion using the SyncAVTM algorithm is superior to CRT with conventional BiV stimulation in the population for which its use is foreseen.

The data will be collected in at least the Selection / Baseline Visit and in the Visit of Follow-up at 6 Months.

The study population are subjects to whom an Abbott Medical CRT has been implanted with SyncAVTM® Stimulation function that go to the participating sites in the study.

The main objective of the study is to assess whether CRT with ventricular stimulation with fusion using the SyncAVTM algorithm is superior to CRT with BiV stimulation conventional in terms of the rate of responders.

The main endpoint is the determination of significant differences between conventional BiV stimulation and ventricular stimulation with fusion using the SyncAVTM algorithm in terms of the percentage of patients responding to CRT therapy with echocardiogram.

The duration of the clinical study is estimated at 24 months with a recruitment period of 18 months and a patient follow-up of 6 months. The number of subjects that is planned to be recruited is 176. The inclusion will be competitive and there is no inclusion number determined per site.

DETAILED DESCRIPTION:
Study design The study is designed post-marketing, prospective, multicenter, randomized and blind for the patient and for the Core-laboratory of the echocardiogram (ECO) department. Has this design is post- marketing since it is a sanitary product with European Committee (CE) marking that is already commercialized and will be used in the study according to its instructions for use. Is a blind study since neither the participant subject nor the Core-laboratory of the ECO (person in charge to assess the main variable of the study) know the treatment that has been randomized the subject, it is a randomized study because the group assignment of each subject is done randomly 1:1.

Study evaluation Evaluation of the risk and benefits of the study: The following will be taking into account

1. Expected clinical benefits:

   * Stimulation function with the SyncAV algorithm is expected increase the rate of responders to therapy.
   * These two methods improve function VI (ventricle left) and it is believed that this additional improvement of the VI function could benefit patients who do not respond to BiV conventional stimulation.
2. Expected adverse effects of the product: bleeding/acute hemorrhage, gas aeration, acceleration of arrythmias, cysts formation, erosion,exacerbation of cardiac insufficiency, venous or cardiac perforation, excessive fibrous tissue development, bruising, histotoxic reactions, infection, keloid formation, myocardial irritability, infection, hematoma, excessive bleeding, local tissue reaction, loss of stimulation and/or detection due to migration or mechanical malfunction, myocardial irritability, stimulation of the nerve, etc. All those events are inherent to the implant of the device for cardiac resynchronization therapy
3. Risk associated with participation in this clinical trial: It is expected that the risks associated with the use of the SyncAVTM stimulation algorithm be comparable to the risks associated with other types of ventricular pacing, and therefore, the risks associated with the use of the stimulation algorithm are expected SyncAVTM will not differ from the risks associated with the different modes of Conventional stimulation available. Patients will be included in the study after the successful implantation of a CRT device, whose indication will be made clinically based on the guidelines current clinical practice of the European Society of Cardiology (ESC).
4. Possible interactions with concomitant medical treatments and / or Simultaneous medical interventions:

No interaction with concomitant pharmacological treatments and / or medical interventions simultaneous, apart from those that occur in the usual treatment with any CRT device. All participants will be candidates for the implantation of a CRT device and will be included in the clinical study once the device has been implanted successfully.

Main Valuation criterion:

The main endpoint of the study is to determine if there are differences significant differences between conventional BiV stimulation and ventricular pacing with fusion using the SyncAVTM algorithm in terms of the percentage of patients responders to CRT therapy

The positive response to CRT is defined as an improvement> 15% in the Systolic Volume End in the Left Ventricle (VSFVI) 6 months after implantation, evaluated by echocardiography.

▪ Secondary rating criterion The secondary endpoints of this study are differences between:

* Inverse remodeling of the VI, measured as the changes in the interval (VTSVI), Volume Telediastolic Left Ventricle (VTDVI), Telesystolic Diameter Left Ventricle (DTSVI), Telediastolic Diaphragm of the Left Ventricle (DTDVI) and Left Ventricular Ejection Fraction (LVEF) at 6 months, in comparison with the Basal situation without stimulation.
* Comparison of the aforementioned echocardiographic parameters with the cohort of patients stratified according to the etiology (ischemic patients versus to non-ischemic patients): or The percentage of super-responder patients * at 6 months. or dyssynchrony measured by the rate of deformation (echocardiography with the speckle tracking technique ) between the anteroseptal segment and the posterior wall (if available). or Electrode position VI: o Short axis (posterolateral, lateral, anterolateral). o Long axis (apical, midventricular, Basal).
* New York Heart Association (NYHA) Class Change at 6 months.
* Mortality from any cause after 6 months.
* Hospitalization rate for any cause, due to cardiovascular causes and / or heart failure, at 6 months.
* Combined mortality and hospitalization variable for heart failure a 6 months
* Quality of life variable according to Kansas City Cardiomyopathy Questionnaire (KCCQ)-12 survey
* % auricular fibrilation (FA) (no patients / FA load)

SAFETY ASSESSMENT The safety of the stimulation algorithms will be evaluated by collecting and registering of any dysfunction, alteration of the features or performance of the product that could or could have led to the death or serious deterioration of the state of health of a patient or a user. Therefore, safety has as an evaluation criterion the Record and analyze the frequency and intensity of adverse incidents that occur throughout the study. For the evaluation of safety, the Population of Security (PS).

Evaluation of effectiveness The superior efficacy of CRT with ventricular stimulation with fusion through SyncAVTM algorithm versus CRT with conventional BiV stimulation will be studied comparing the results of the stimulation logarithms between the two branches of the study (stimulation by SyncAVTM algorithm and conventional BiV stimulation).The ultimate goal of the study is to determine the percentage of responding patients and not respondents The response of patients to CRT will be evaluated taking into account the reduction of VSFVI. Patients will be classified as responders. have documented a reduction in VSFVI of at least 15% compared to the data collected in the Basal situation without stimulation. The evaluation of the effectiveness will be analyzed with the Population of Intent to Treat (ITT) and Population by Protocol (PP).

Sample size The calculation of the sample size is based on the main variable: the proportion of responders to CRT at 6 months with the SyncAV function activated at the start of the study.

The main variable of the study is the response to re-synchronization, understood as a dichotomous variable that takes the values: Yes / No. In the study there will be two randomization groups, and the response rate of the control group is set at 65% of the patients, while that of the study group will be 77%, that is, 12% higher. As statistical criteria for the estimation of the sample size, it was used a confidence level of 95%, a margin of non-inferiority δ = 0 and a power a priori of 80%. The statistical technique used for the analysis of the main variable is a test χ 2

The formula used to calculate the sample size is as follows (Chow, Shao and Wang, 2008): In addition, it is assumed that 5% of patients may be lost due to loss of follow-up and 8% due to exitus. For the calculation of the sample size, the R-studio software (version 1.0.153). Applying the formula, the sample size is 77 patients per group, that is, a total of 154 patients. However, 22 more must be added (11 more patients in each group) due to possible loss of follow-up and due to death.

Considering all the above information, the expected sample size is of 176 patients, 88 patients would be randomized to the control group and 88 to the group of study.

Using an exact binomial test of a unilateral sample, with a level of significance of 95%, a total of 176 patients would be necessary to reach a 80% power.

To detect a difference of 12% between the two responder rates, it is It is necessary that a total of 176 patients have analysable data at 6 months.

Based on clinical experience, it is assumed that some patients will abandon the study (5% during the first 6 months of implantation, 8% due to exitus)

STATISTICAL ANALYSIS

Statistical design, hypothesis, method and analytical procedures:

The analysis of the main variable will be based on the intention to treat principle (ITT), including all deviations from the Protocol. There will also be a secondary analysis per Protocol (PP), excluding all deviations of the Protocol. If the results obtained in these analyzes were different, an exploration of the data will be done in search of the reasons. In the analysis of the main variable will be evaluated the following hypothesis of inequality:

* H0: Proportion of responders at 6 months with ventricular stimulation with fusion using SyncAVTM algorithm <Proportion ofResponders at 6 months with conventional BiV stimulation.
* H1: Proportion of responders at 6 months with ventricular stimulation with fusion using the SyncAVTM algorithm > Proportion ofResponders at 6 months with conventional BiV stimulation.

All results will be expressed according to the corresponding intervals confidence of 97.5% and the values p. P values less than 2.5% are will consider significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients who state that they understand the study and are willing to participate in it by signing the corresponding Informed Consent form.
* Patients who have been implanted with an Abbott Medical ® CRT with SyncAVTM stimulation function under the current ESC Class I or Class II-a indications for the implantation of CRT (including updates from pacemakers or single-chamber or double-chamber of an implantable cardioverter-defibrillator (ICDs)).
* In sinus rhythm during the Basal visit.
* Patients with Left Branch Block (LBB) defined as:

  * QRS duration> 120 msec
  * interval (QS) or interval (rS) in V1
  * Single phase R (without Q wave) in V6 and interval (DI)
* LVEF <35% being under optimal medical treatment
* PR Baseline <250 ms without BAV of 2nd or 3rd grade.
* Patients who are willing to meet all the requirements of the study and who have the ability to do it.

Exclusion Criteria:

* Having suffered myocardial infarction or unstable angina in the 40 days prior to inclusion.
* NYHA Class IV.
* Having undergone coronary revascularization (PTCA, Stent or CABG) in the 4 weeks prior to inclusion.
* Having suffered a cerebrovascular accident (CVA) or a Transient Ischemic Accident (TIA) in the 3 months prior to inclusion.
* Have a status of 1 for heart transplantation or be evaluated to receive a transplant in the next 12 months.
* Primary valve disease that requires surgical intervention.
* 2nd or 3rd grade of AV block.
* PR> 250 ms.
* Atrial Fibrillation (AF): Persistent AF at the time of inclusion or 30 days before, or permanent FA not treated with ablation of the AV node in the 2 weeks following the implantation of the CRT, or History or incidence of Paroxysmal or Persistent FA in the 30 days prior to inclusion.
* Patient in whom adequate transthoracic echocardiographic images can not be obtained to establish cardiac output and VI volumes.
* Have received a heart transplant or are waiting to receive it.
* Have a life expectancy <6 months.
* Being pregnant or intending to become pregnant during the study.
* Inability to comply with the follow-up calendar.
* Being currently participating in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Number of responders patients evaluating the superiority of CRT with ventricular stimulation with fusion using the SyncAV TM algorithm versus BiV conventional stimulation | 6 months
  The assessment of the main objective must be carried out on a population that has been implanted an Abbott Medical® CRT with SyncAV TM Stimulation function under the current ESC Class I or Class II-a indications for CRT implantation (including pacemaker or single-chamber or dual chamber of an implantable cardioverter defibrillator (DAI) updates

SECONDARY OUTCOMES:
Inverse remodeling of the LV | 6 months
  It will be measured as the changes into the left ventricle end systolic volume (LVESV) and left ventricle end diastolic volume(LVEDV) in comparison with the Basal situation without stimulation.
  Changes of LV will be measured by echocardiogram in the apical 4-chamber plane using General Electric equipment (VIVID E9) and reviewing images obtained by VIVID E9 program following the GUIDELINES AND STANDARDS "Recommendations for Cardiac Chamber Quantification by Echocardiography in Adults: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging".
Inverse remodeling of the LV | 6 months
  It will be measured as the changes into the Left Ventricle end diastolic diameter (LVEDD) in comparison with the Basal situation without stimulation.
  Changes of LV will be measured by echocardiogram in the apical 4-chamber plane using General Electric equipment (VIVID E9) and reviewing images obtained by VIVID E9 program following the GUIDELINES AND STANDARDS "Recommendations for Cardiac Chamber Quantification by Echocardiography in Adults: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging".
Inverse remodeling of the LV | 6 months
  It will be measured as the changes into the Left Ventricular Ejection Fraction (LVEF) in comparison with the Basal situation without stimulation.
  Changes of LV will be measured by echocardiogram in the apical 4-chamber plane using General Electric equipment (VIVID E9) and reviewing images obtained by VIVID E9 program following the GUIDELINES AND STANDARDS "Recommendations for Cardiac Chamber Quantification by Echocardiography in Adults: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging"
Quality of life variable according to KCCQ-12 survey | 6 months
  It comprises 23 items in seven domains: physical limitation; symptoms, with domains for change over time, frequency, and severity; self-efficacy and knowledge; quality of life; and social interference. The response options for the items are Likert-type scales ranging from 1 to 5, 6 or 7 points and the score on each domain can, in theory, range from 0 to 100, with 100 corresponding to the best state
Number of appropriate / inappropriate discharge in patients | 6 months
  Throughout the visits dates and/or hospital incoming.
% of patients with AF and AF load | 6 months
  These % of Atrial fibrilation will be evaluated by each MD at the site face-to-face with the patients.
% of patients who lose the possibility of SyncAV TM (BAV, lengthening of interval (PR) ...) | 6 months
  Throughout the visits dates and/or hospital incoming.
Comparison of the echocardiographic parameters with the cohort of patients stratified according to the etiology (ischemic patients versus to non-ischemic patients) | 6 months
  Comparison of the echocardiographic parameters with the cohort of patients stratified according to the etiology (ischemic patients versus to non-ischemic patients)
NYHA Class Change | 6 months
  By evaluating it at the on-site visit from each patients
Mortality from any cause | 6 months
  Mortality from any cause
Hospitalization rate for any cause, due to cardiovascular causes and / or heart failure | 6 months
  Hospitalization rate for any cause, due to cardiovascular causes and / or heart failure
Combined mortality and hospitalization variable for heart failure | 6 months
  Combined mortality and hospitalization variable for heart failure
% FA (no patients / FA load) | 6 months
  % FA (no patients / FA load)

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Francisco Pascual, MD, Principal Investigator — Institut of research Vall d'hebron Hospital (VHIR)
Locations (15):
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Insular de las Palmas, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario Puerta del Mar, Cadiz, Vizcaya
  - Hospital Universitario de Galdakao, Galdakao, Vizcaya
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Girona Dr. Josep Trueta, Girona
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital Álvaro Cunqueriro, Pontevedra
  - Hospital Virgen de la Salud, Toledo
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared to other researchers.